CLINICAL TRIAL: NCT06065839
Title: Effect of Non-nutritive Sucking on Feeding Intolerance in Premature Infants
Brief Title: Effect of Non-nutritive Sucking on Feeding Intolerance
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, HUANG, YU-TING, Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 202201089A3
Record Dates: First submitted 2023-09-03; First posted 2023-10-04 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Non-nutritive Sucking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): non-nutritive sucking was not given before feeding
- Experimental group A (Active Comparator): Give pacifier non-nutritive sucking for 5 minutes before feeding
  Interventions: Other: non-nutritive sucking 5 minutes
- Experimental group B (Placebo Comparator): Give pacifier non-nutritive sucking for 15 minutes before feeding
  Interventions: Other: non-nutritive sucking 15 minutes

INTERVENTIONS:
Other: non-nutritive sucking 5 minutes — Give pacifier non-nutritive sucking for 5 minutes before feeding
  Arms: Experimental group A
Other: non-nutritive sucking 15 minutes — Give pacifier non-nutritive sucking for 15 minutes before feeding
  Arms: Experimental group B

SUMMARY:
The design of this study is an experimental research design, and the research subjects who meet the conditions of acceptance will be used as randomized controlled trials. Cases meeting the sampling conditions in the neonatal intensive care unit were stratified according to birth weeks (26 to 27+6 weeks and 28 to 31+6 weeks), and then randomly assigned to experimental group A (non-nutritive sucking 5 minutes), experimental group B (non-nutritive sucking for 15 minutes) and control group (no non-nutritive sucking). The variables controlled in this study were gestational weeks, birth weight, sex, Apgar score, respirator use, and type of milk fed. The premature infants in the experimental group were given non-nutritive sucking before the first tube-feeding and the feeding volume reached 10mL/kg/day, while the control group was not given non-nutritive sucking before tube-feeding.

The interventional measures adopted in this study were set as two meals a day before 17:00, and the patients were force-fed every three hours, and the time interval between the two interventional measures was every six hours (intervention measures were provided every other meal) , the measurement time, times and intervals of the two groups are the same. Experimental group A was given pacifier NNS 5 minutes before each feeding, experimental group B was given pacifier NNS 15 minutes before each feeding, while the control group was not given NNS before feeding, and the two groups were given 150 minutes after feeding (ie 30 minutes before the next force-feeding) to monitor gastric residual volume, changes in abdominal circumference, and vomiting. Since FI mainly occurred 48-72 hours after the start of feeding, the duration of this study was 3 consecutive days to compare with the control group.

The acceptance conditions of the research objects are: 1. Premature infants whose gestational age is more than 26 weeks (inclusive) to less than 32 weeks, 2. Premature neonates who have been placed with orogastric tube or nasogastric tube for force-feeding, 3. No congenital gastrointestinal tract Abnormal, 4. No serious congenital abnormalities and heart disease, no cleft lip and palate, 5. Never received stomach or intestinal surgery, 6. No central nervous system damage, 7. With the consent of their parents or guardians, and fill out the consent form By. If the condition is unstable during the course of the case, including severe hypoxemia, hypotension, esophageal perforation, necrotic enteritis, sepsis caused by infection, and grade 3-4 intraventricular hemorrhage, etc., they will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Premature infants whose gestational age is more than 26 weeks (inclusive) to less than 32 weeks
* Premature neonates who are force-fed with orogastric or nasogastric tubes
* No congenital gastrointestinal abnormalities
* No serious Congenital anomalies and heart disease, no cleft lip and palate
* Never received stomach or intestinal surgery
* No central nervous system damage
* With the consent of their parents or guardians, and fill out the consent form.

Exclusion Criteria:

* Severe hypoxemia
* Severe hypotension
* Esophageal perforation
* Necrotic enteritis
* Infection-induced sepsis
* 3-4 grades of ventricular hemorrhage

Ages: 26 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Estimated)
Dates: Start 2022-09-20 (Actual); Primary Completion 2024-08-16 (Estimated); Study Completion 2024-08-16 (Estimated)

PRIMARY OUTCOMES:
feeding intolerance | The test was carried out twice a day, with an interval of 6 hours between each data collection, and the test was carried out continuously for 3 days
  Gastric residual volume in milliliter
feeding intolerance | The test was carried out twice a day, with an interval of 6 hours between each data collection, and the test was carried out continuously for 3 days
  abdominal circumference in centimeter
feeding intolerance | The test was carried out twice a day, with an interval of 6 hours between each data collection, and the test was carried out continuously for 3 days
  vomiting in frequency

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Ting HUANG, BSN, Principal Investigator — Chang Gung Memorial Hospital; Shi-Fang TSENG, BSN, Study Chair — Chang Gung Memorial Hospital; Jian-Tao LEE, PhD, Study Director — Chang Gung University
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Kwei-Shan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bernbaum JC, Pereira GR, Watkins JB, Peckham GJ. Nonnutritive sucking during gavage feeding enhances growth and maturation in premature infants. Pediatrics. 1983 Jan;71(1):41-5. PMID 6401358
- [Background] Szabo JS, Hillemeier AC, Oh W. Effect of non-nutritive and nutritive suck on gastric emptying in premature infants. J Pediatr Gastroenterol Nutr. 1985 Jun;4(3):348-51. doi: 10.1097/00005176-198506000-00004. PMID 4020566
- [Result] Foster JP, Psaila K, Patterson T. Non-nutritive sucking for increasing physiologic stability and nutrition in preterm infants. Cochrane Database Syst Rev. 2016 Oct 4;10(10):CD001071. doi: 10.1002/14651858.CD001071.pub3. PMID 27699765
- [Result] Marchini G, Lagercrantz H, Feuerberg Y, Winberg J, Uvnas-Moberg K. The effect of non-nutritive sucking on plasma insulin, gastrin, and somatostatin levels in infants. Acta Paediatr Scand. 1987 Jul;76(4):573-8. doi: 10.1111/j.1651-2227.1987.tb10523.x. PMID 2888258
- [Result] Widstrom AM, Marchini G, Matthiesen AS, Werner S, Winberg J, Uvnas-Moberg K. Nonnutritive sucking in tube-fed preterm infants: effects on gastric motility and gastric contents of somatostatin. J Pediatr Gastroenterol Nutr. 1988 Jul-Aug;7(4):517-23. doi: 10.1097/00005176-198807000-00007. PMID 2899621

DOCUMENTS (1):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT06065839/Prot_000.pdf